CLINICAL TRIAL: NCT02228707
Title: A Randomized, Double-Blind, Placebo-Controlled, Multiple Ascending Dose Study of the Safety, Tolerability, and Pharmacokinetics of BIIB061 in Healthy Adult Volunteers
Brief Title: Study to Assess the Safety, Tolerability, and Pharmacokinetics of BIIB061 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 231HV102
Record Dates: First submitted 2014-08-27; First posted 2014-08-29 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BIIB061 (Experimental): Participants receive BIIB061
  Interventions: Drug: BIIB061
- Placebo (Placebo Comparator): Participants receive matched placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BIIB061 — Participants receive BIIB061
  Arms: BIIB061
Other: Placebo — Matched placebo
  Arms: Placebo

SUMMARY:
The primary objectives of the study are to evaluate the safety and tolerability of multiple doses of BIIB061 administered to healthy adults. The secondary objective is to determine the multiple-dose PK profile of BIIB061 in this study population.

ELIGIBILITY:
Key Inclusion Criteria:

* Males and postmenopausal (defined as no menses for 12 months and confirmed by follicle-stimulating hormone [FSH] levels determined at screening to be in the postmenopausal range) or surgically sterile females
* Must be in good health and have normal vital signs as determined by the Investigator, based on medical history and screening evaluations.
* Must agree to abstain from alcohol ingestion for the duration of the study.
* Must agree to abstain from consumption of grapefruit or grapefruit-containing products for the duration of the study, starting at least 24 hours prior to admission to the inpatient facility.
* Must agree to abstain from taking St. John's Wort (herbal preparation) for the duration of the study
* Must agree to abstain from any vigorous exercise (as determined by the Investigator) for the duration of the study.
* Must have a body mass index of 18 to 30 kg/m2, inclusive.

Key Exclusion Criteria:

* History of or positive test result at screening for human immunodeficiency virus, hepatitis C virus antibody, or hepatitis B virus (defined as positive for hepatitis B surface antigen [HBsAg] or hepatitis B core antibody [HBcAb]).
* Presence of a metal device (e.g., any type of electronic, mechanical, or magnetic implant; cardiac pacemaker; aneurysm clips; implanted cardiac defibrillator) or potential ferromagnetic foreign body (metal slivers, metal shavings, other metal objects) that are contraindications for MRI.
* History of asthma, wheezing, allergies involving the lungs, or airway obstruction.
* History of bronchodilator or inhaler use.
* Clinically significant abnormal hematology or blood chemistry values, as determined by the Investigator.
* Inability or unwillingness to comply with study requirements.
* Other unspecified reasons that, in the opinion of the Investigator or Biogen Idec, make the subject unsuitable for enrollment.

Note: Other protocol defined inclusion/ exclusion criteria may apply.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Number of participants experiencing AEs | Up to 28 days post treatment period (Day 1 to Day 56)

SECONDARY OUTCOMES:
Plasma BIIB061 Concentration | Up to 28 days post treatment period (Day 1 to Day 56)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Madison, Wisconsin, United States